CLINICAL TRIAL: NCT02059109
Title: Evaluation of a Training Model for the Proficient Use of the Belmont Rapid Infuser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2011-1844
Record Dates: First submitted 2014-01-29; First posted 2014-02-11 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Use of the Belmont Rapid Infuser
Keywords: Belmont; Rapid; Infuser; proficiency; proficient; training
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single (Experimental): Staff will work alone to assemble the Belmont Rapid Infuser
  Interventions: Procedure: Hands on Assembly of Belmont Rapid Infuser
- Pair (Experimental): Staff will work in pairs to assemble the Belmont Rapid Infuser
  Interventions: Procedure: Hands on Assembly of Belmont Rapid Infuser

INTERVENTIONS:
Procedure: Hands on Assembly of Belmont Rapid Infuser — Participants will work individually or in pairs to assemble the Belmont Rapid Infuser in addition to completing the traditional training methods.

SUMMARY:
The Belmont Rapid Infuser is a device currently approved to replace larger volumes of necessary fluids such as blood in a fast and safe manner. The purpose of the study is to evaluate proficiency and the retention of knowledge of how to use the device based on current methods of training compared to revised training methods.

Hypotheses:

1. The use of the traditional method of training is not effective, predicting less then half of staff will pass on the first attempt.
2. Restructured test with hands-on training as opposed to oral presentation only with a written test will result in a pass rate of > 80%.
3. Staff members who work in pairs will perform better than working alone when setting up the Belmont Rapid Infuser (BRI).
4. Retention at 3 months will be higher with the restructured training method than with the traditional training method.

DETAILED DESCRIPTION:
Participants will be recruited to complete a test after undergoing either the traditional or the restructured training method. This training will be completed on one day and takes about 1 hour.

All participants who pass via either method of training are evaluated again to test retention 3-4 months later .

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited from the faculty, Certified Registered Nurse Anesthetists, and fellows from the Department of Anesthesia at Cincinnati Children's Hospital Medical Center.
* They may have had educational exposure or use of the Belmont Rapid Infuser without independent assembly.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Proficiency | Measured after the training session (approximately 1 hour).
  The composite score of "pass-pass" on BRI assembly and on knowledge test .

SECONDARY OUTCOMES:
Retention of proficiency | 3 -4 months after delivery of the effective teaching model.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Medical Center, Cincinnati, Ohio, United States